CLINICAL TRIAL: NCT04590456
Title: Efficacy of Pulsed Electromagnetic Field on Hemarthrotic Knee in Haemophilic Adolescence
Brief Title: Pulsed Electromagentic Field in Haemophilia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, walaa eldesoukey heneidy, lecturer of physical therapy, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEMF
Record Dates: First submitted 2020-09-22; First posted 2020-10-19 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Experimental)
  Interventions: Other: PEMF
- PEMF group (Experimental)
  Interventions: Other: PEMF

INTERVENTIONS:
Other: PEMF — group A received 60 minutes of traditional program physical therapy which consisted of passive range of motion, stretching,proprioception, isotonic and isometric and 20 minutes of placebo treatment using PEMF, while group B received the same traditional physical therapy program given to the control group in addition of 20 minutes of PEMF therapy

SUMMARY:
To assess the effect of pulsed electero- magnetic field on swelling, range of motion and muscle strength of hemarthrotic knee joints of haemophilic subjects.

DETAILED DESCRIPTION:
Haemophilia is an X-linked hereditary sex recessive disorder that impairs the body's ability to make blood clots. It includes two types: A (FVIII deficit factor) and B (IX deficit factor), depending on FVIII/FIX percentage in blood. The severity of haemophilia is classified into (severe: <1%, moderate: 1-5%, and mild: >5%). The prevalence of haemophilia A is 1: 5000 live births and haemophilia B is 1: 30000 live births.

This disease is characterized by hemarthrosis which is a hemorrhage in the locomotor system, mainly muscles and joints. Joint bleeding mainly occurs in knees, ankles and elbows. Haemorrhage in the muscle or joints accounts for 80% to 90% of all bleeding episodes in people with haemophilia. The most commonly affected joints in non-prophylaxis patients are the knees (45%) which is thought to be due to the large size of the synovial membrane and large rotational forces present. It is followed by the elbows (30%), ankles (15%), shoulders (3%), and wrists (2%). Bleeds are best detected by the patients themselves as bruising and swelling or described as a feeling of warmth or tingling within the joint preceding the clinical signs.

Pulsed electromagnetic field (PEMF) has been reported to be effective in reducing pain, healing of ulcers and promote bone healing, and treating osteoarthritis and inflammatory diseases of the musculoskeletal system. Also, it was reported that PEMF exposure significantly increases the anti-inflammatory effect, suggesting its potential therapeutic use in the treatment of inflammatory bone and joint disorders.

ELIGIBILITY:
Inclusion Criteria:

* type A hemophilia (moderate)
* free from any musculoskeletal deformities.

Exclusion Criteria:

* patients who performed surgical procedures 6 weeks before conducting the study

Ages: 13 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-19 (Estimated); Study Completion 2020-12-19 (Estimated)

PRIMARY OUTCOMES:
swelling | basline and after 3 months of intervention.
  The swelling degree was detected by tape

SECONDARY OUTCOMES:
range of motion | basline and after 3 months of intervention.
  Active knee range of flexion and extension were measured by electronic goniometer.
muscle strength | basline and after 3 months of intervention.
  The peak concentric knee extensor (KE) and the peak concentric knee flexor (KF) was measured at 60/s angular speed by an isokinetic dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Hala I. Kassem, Professor, Study Chair — Professor of physical therapy
Locations (1):
- Delta University for Science and Technology, Gamasa, Dakahelia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gringeri A, Ewenstein B, Reininger A. The burden of bleeding in haemophilia: is one bleed too many? Haemophilia. 2014 Jul;20(4):459-63. doi: 10.1111/hae.12375. Epub 2014 Jan 29. PMID 24472015